CLINICAL TRIAL: NCT04889287
Title: Open-label, One-sequence Crossover Study to Determine the Effects of Multiple Doses of Elinzanetant on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Brief Title: A Study to Learn How Much Rosuvastatin Gets Into the Blood When Taken With or Without Elinzanetant and to Learn About the Safety of Elinzanetant in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 21666; 2020-004635-25 (EudraCT Number)
Record Dates: First submitted 2021-05-14; First posted 2021-05-17 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men
Keywords: Vasomotor symptoms
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin and/or elinzanetant (Experimental): The participants will receive each dose of rosuvastatin and/or elinzanetant together with 240 mL of non-sparkling water in total.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Rosuvastatin

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Once daily over 12 days
Drug: Rosuvastatin — Single doses on Day 1, Day 8, and Day 13

SUMMARY:
Researchers are looking for a better way to treat people who have symptoms caused by hormonal changes, like those that happen in women during menopause. These symptoms can include vasomotor symptoms. Before a treatment can be approved for patients to take, researchers do clinical studies to better understand its safety and what happens to the treatment in the body.

The study drug, elinzanetant, was designed to treat vasomotor symptoms. Rosuvastatin is already approved for doctors to prescribe and is used to treat high cholesterol levels and prevent heart problems. It is important for researchers to know if taking elinzanetant will affect how other drugs work in the body. Researchers regularly use rosuvastatin in studies to learn how it affects drugs like elinzanetant.In this study, the researchers will study how much elinzanetant gets into the participants' blood when taken with or without rosuvastatin. The study will include about 16 male participants who are between 18 and 65 years old. The participants will all take 5 milligrams (mg) of rosuvastatin and 120 mg of elinzanetant as capsules by mouth. On some days, they will take only rosuvastatin or only elinzanetant. On other days, they will take both study treatments. Each participant will be in the study for up to 6 weeks. But, the entire study will last about 2.5 months.

During the study, all of the participants will stay at the study site for 17 days. Blood and urine samples will be collected. The physician will also check the participants' heart health using an electrocardiogram (ECG). The participants will answer questions about how their well being and taken medications.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG, vital signs, respiratory rate and body temperature.Weight.
* Body weight above or equal 50 kg and body mass index (BMI) within the range 18.0 and 30.0 kg/m*2 (inclusive).
* Male.
* Contraceptive use by men or female partners of male participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

  -- a. Male participants:
  * Male participants of reproductive potential must agree to use a condom (with or without spermicide) when sexually active. This applies for the time period between the signing of the informed consent form until 7 days after the last dose of study intervention.
  * Female partners of childbearing potential of male participants do not need to follow special precautions.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* History or evidence of any clinically relevant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other clinically relevant disease, as judged by the investigator.
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal.
* Use of any systemic or topical medicines or substances which oppose the study objectives, or which might influence them (for further information, see Section 6.8) within 4 weeks prior to screening.
* Participants with positive serology for any of hepatitis B, hepatitis C, of HIV.
* Clinically relevant deviations of the screened safety laboratory parameters in clinical chemistry, hematology, or urinalysis from reference ranges.
* Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular (AV) block, prolongation of the QRS complex over 120 msec or QT interval frequency-corrected according to Bazett's formula (QTcB) -prolongation over 450 msec at screening.
* Participants with a presence of any of the following, confirmed by a repeat test: AST, alanine aminotransferase (ALT) and/or bilirubin above 1.2 x upper limit of normal (ULN) (at screening or Day -1).
* Known intolerance to statins.
* Current or medical history of myopathy, rhabdomyolysis or myasthenia.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of rosuvastatin when given without or together with elinzanetant | Day 1-3, Day 8-16
Area under the concentration versus time curve (AUC) of rosuvastatin when given without or together with elinzanetant | Day 1-3, Day 8-16

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Approximately 2.5 months
Severity of treatment-emergent adverse events (TEAEs) | Approximately 2.5 months

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.